CLINICAL TRIAL: NCT01805440
Title: Placebo-Controlled Study of Uridine for Adolescent Bipolar Depression: a Magnetic Resonance Spectroscopy Study
Brief Title: Uridine Adolescent Bipolar Depression Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Douglas Kondo, MD, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: University of Utah
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Bipolar Disorder; Bipolar Depression; Manic Depression
Keywords: Adolescent; Bipolar Disorder; Bipolar Depression; Manic Depression; Neuroimaging; Magnetic Resonance Spectroscopy; Uridine; Pyrimidines
MeSH Terms: conditions — Bipolar Disorder | interventions — Uridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Uridine (Active Comparator): Subjects randomized to this study arm will receive uridine 500 mg twice daily by mouth for 6 weeks.
  Interventions: Drug: Uridine
- Placebo (Placebo Comparator): Subjects randomized to this arm of the study will receive placebo 500 mg twice daily by mouth for 6 weeks.
  Interventions: Drug: Placebo
- Healthy Comparison (No Intervention): Subjects are not randomized, and do not receive any treatment intervention.

INTERVENTIONS:
Drug: Uridine — Uridine is the active treatment in this clinical trial.
  Arms: Uridine
Drug: Placebo — Pill placebo is the inactive treatment comparator in this clinical trial.
  Other Names: Pill Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of the investigational drug uridine as a treatment for depressed adolescents with bipolar disorder (i.e. "bipolar depression"). Participants initially randomized to placebo who complete the 6-week protocol will be offered 6 months of open-label uridine treatment and follow-up. Participants initially randomized to uridine will be offered the open-label treatment as well.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of the investigational drug uridine as a treatment for depressed adolescents with bipolar disorder (i.e. "bipolar depression").

In addition to treatment with the investigational drug versus placebo, the study includes a translational neuroimaging component: magnetic resonance spectroscopy (1H-MRS) brain scans are performed at baseline, and then repeated following 6 weeks of treatment with uridine or placebo. The scans do not use radiation, and are performed on a 3 Tesla MRI system that is approved for clinical use. The scans allow researchers to measure the concentrations of several chemicals in the brain that are believed to be involved in bipolar disorder and depression.

The primary hypothesis is that uridine treatment will be associated with a significant decrease in GLX (i.e. glutamate + glutamine) levels, compared to placebo, in a part of the brain known as the anterior cingulate cortex.

The secondary hypothesis is that decreased depressive symptoms measured with the Children Depression Rating Scale-Revised (CDRS-R) and Montgomery-Asberg Depression Rating Scale (MADRS) will be correlated with reductions in GLX.

All participants who complete the initial 6-week protocol, including two brain scans, will be offered 6 months of open-label treatment with uridine.

ELIGIBILITY:
Inclusion Criteria For Bipolar Disorder Participants:

* Participants under 18 years of age must be able to provide assent, and have the permission of a parent or guardian. Participants 18 years of age or older must be able to provide informed consent.
* Participants must be between the ages of 13 and 21 years.
* Participants must meet DSM criteria for Bipolar Disorder (Type I, II, or NOS), with current mood state depressed for at least 2 weeks.
* Participants must have a current Children's Depression Rating Scale-Revised (CDRS-R) score of 45 or greater, and/or a Montgomery/Asberg Depression Rating Scale (MADRS) score of 25 or greater.

Inclusion Criteria For Healthy Comparison Participants:

* Participants under 18 years of age must be able to provide assent, and have the permission of a parent or guardian. Participants 18 years of age or older must be able to provide informed consent.
* Participants must be between the ages of 13 and 21 years.
* Participants must not meet any DSM-IV criteria for a psychiatric illness or substance use disorder

Exclusion Criteria:

* Participants must not meet DSM criteria for a primary psychotic disorder, a developmental disorder or substance use disorder.
* Participants must not be at high risk for suicidal or homicidal actions.
* Participants must not be pregnant or breastfeeding.
* Participants must not have a contraindication to magnetic resonance imaging (e.g. ferromagnetic implant, or claustrophobic anxiety).
* Incarcerated persons are excluded, because this study is not approved for Research Involving Prisoners.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondo, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Informed Consent to publicly share individual participant data, e.g. MRI and MRS brain scans, was not obtained.

REFERENCES:
- [Background] Kondo DG, Sung YH, Hellem TL, Delmastro KK, Jeong EK, Kim N, Shi X, Renshaw PF. Open-label uridine for treatment of depressed adolescents with bipolar disorder. J Child Adolesc Psychopharmacol. 2011 Apr;21(2):171-5. doi: 10.1089/cap.2010.0054. Epub 2011 Apr 12. PMID 21486171
- See also: Free downloadable full-text article — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3080753/

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Comparison: Subjects seen for screening and baseline scan. No randomization or treatment intervention for subjects enrolled as a Healthy Comparison.
Period: Overall Study
Arm/Group | Uridine | Placebo | Healthy Comparison
Started | 19 | 17 | 26
Completed | 18 | 17 | 26
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uridine | Placebo | Healthy Comparison | Total
Number analyzed (Participants) | 19 | 17 | 26 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 6 | 22
  Between 18 and 65 years | 9 | 11 | 20 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.74 (2.28) | 18.29 (2.62) | 18.54 (2.37) | 17.47 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 16 | 40
  Male | 5 | 7 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in GLX (Glutamate + Glutamine) to Creatine (Cr) Ratio in the Anterior Cingulate Cortex of the Brain, as Measured With Proton-1 Magnetic Resonance Spectroscopy (1H-MRS).
Description: Magnetic Resonance Spectroscopy is a safe, non-invasive method for measuring brain chemicals thought to be involved in mood disorders, such as GLX (glutamate + glutamine). Previous research indicates that adolescents with bipolar depression have elevated Glx concentrations, compared with controls. The measurement of Glx with 1H-MRS has the potential to identify translational biomarkers of juvenile BD pathophysiology and treatment response.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Brain GLX/Cr
Groups:
- Healthy Comparison: Subjects did not receive study medication. Subjects were only seen for baseline visit.
Arm/Group | Uridine | Placebo | Healthy Comparison
Number analyzed (Participants) | 18 | 17 | 26
Brain GLX/Cr
  Before treatment | 1.5731 (.1082) | 1.6557 (.1105) | 1.6051 (.1195)
  After 6 weeks treatment | 1.6738 (.1147) | 1.6121 (.0977) | NA (NA) — Subjects were healthy comparisons, and were only seen once at baseline.

2. Primary Outcome: Change in Children's Depression Rating Scale-Revised (CDRS-R) Score.
Description: The CDRS-R is a brief rating scale based on a semi-structured interview with the participant (and/or their parent or guardian). The scale can be administered and scored in under 30 minutes. The CDRS-R gives you a single summary score -- with an interpretation of, and clinical recommendations for, six different score ranges. Total possible scores range from 17 to 113, with higher scores indicating more depressive symptoms reported by the participant (and/or their parent or guardian).
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Uridine | Placebo | Healthy Comparison
Number analyzed (Participants) | 18 | 17 | 26
Units on a scale
  Total Score before treatment | 59.05 [49 to 74] | 58.18 [43 to 74] | 21.31 [17 to 28]
  Total Score after 6 weeks treatment | 45.67 [30 to 74] | 36.76 [21 to 64] | NA [NA to NA] — Subjects were healthy comparisons, and were only seen once at baseline.

3. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is used to measure suicidal thoughts and behaviors in Investigational New Drug (IND) studies. The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Uridine | Placebo | Healthy Comparison
Number analyzed (Participants) | 18 | 17 | 26
Scores on a Scale
  Participants SI Severity at Baseline | 0.6875 (0.7932) | 0.5882 (1.0690) | 0 (0)
  Participants SI Severity after 6 Weeks Treatment | 0.5 (0.6183) | 0.4706 (1.0676) | NA (NA) — Subjects were healthy comparisons, and were only seen once at baseline.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants at every visit, starting after the treatment intervention was dispensed at baseline. Adverse events were assessed up to 6 weeks.
Description: Healthy comparison participants were only seen at baseline, and were not exposed to any treatment intervention, therefore, adverse events were not collected.
Arm/Group | Uridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/17
Other Adverse Events (participants affected / at risk) | 12/19 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uridine (N=19) | Placebo (N=17)
Other Serious (Important Medical Event) (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uridine (N=19) | Placebo (N=17)
Stomach Discomfort (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 5 | 3

LIMITATIONS AND CAVEATS:
Limited sample size and small percentage of underrepresented racial/ethnic minority participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No